CLINICAL TRIAL: NCT06827197
Title: Role of Interleukin-1β and Prostaglandin E2 in Prediction and Outcome of Apnea in Neonates
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amany Mohammed El-Rebigi, MD, Lecturer of Pediatrics, Faculty of Medicine, Benha University, Benha, Egypt, Benha University
Other Study IDs: MS 4-5-2023
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Premature Newborns; Premature Newborns With Gestational Age 28 to 33 Weeks
Keywords: Apnea of prematurity; Interleukin-1β; Prostaglandin E2; Outcome
MeSH Terms: conditions — Apnea | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood test — Blood samples were withdrawn from all the neonates under strict aseptic conditions and stored at -80°C for detecting PGE2 and IL-1β levels. PGE2 and IL-1β concentrations were measured using ELISA.

SUMMARY:
Our thesis proposed that IL-1β may affect brainstem respiratory control via prostaglandin-dependant mechanism so we investigated the mediator roles of IL-1β and PGE2 levels in predicting apnea in pretertm newborn and their relation to clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at less than 37 weeks of gestation.
* Neonates aged from birth up to 28 days.
* Neonates diagnosed with apnea of prematurity or exhibiting apneic episodes

Exclusion Criteria:

* Full-term neonates.
* Neonates with major congenital malformations or genetic syndromes.
* Neonates with severe neurological impairments (e.g., intraventricular hemorrhage grade III or IV).
* Neonates with confirmed or suspected sepsis or active infections.
* Neonates receiving steroids, nonsteroidal anti-inflammatory drugs (NSAIDs), or other medications known to alter interleukin-1β or prostaglandin E2 levels.
* Neonates with congenital heart diseases.
* Neonates with a history of significant birth asphyxia requiring extensive resuscitation.
* Neonates whose parents or guardians refuse to provide informed consent.

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study included 100 preterm neonates who were recruited from the Neonatal Intensive Care Unit, Pediatric Department of Benha University Hospital, during the period from May 2023 till October 2023. They were eligible for the study and their parents agreed to participate in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Duration of NICU stay | 1 month
Mortality rate | 1 month

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Benha University, Cairo, Al-Qalyubia
  - Amany El-Rebigi, Banhā

IPD SHARING:
Plan to Share IPD: No